CLINICAL TRIAL: NCT00810823
Title: The Effect of Gastric Bypass Surgery on the Glucose Metabolism Seen in Patients With Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Professor, DMSc Sten Madsbad, Hvidovre Univesity Hospital, department of endocrinology
Other Study IDs: H-A-2008-080
Record Dates: First submitted 2008-12-17; First posted 2008-12-18 (Estimated); Last update posted 2011-07-06 (Estimated); Status verified 2008-12

CONDITIONS: Type 2 Diabetes
Keywords: Diabetes; gastric bypass; type 2 diabetes and gastric bypass
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1:Gastric bypass/diabetes: Patients undergoing gastric bypass surgery, and who are diagnosed with type 2 diabetes.
- 2:Gastric bypass/not Diabetic: Patients undergoing gastric bypass surgery, not diagnosed with diabetes.

SUMMARY:
Gastric bypass surgery has in many studies shown total remission of type 2 diabetes as early as 1 - 2 days after surgery and this is before any real weight loss has occurred. This suggest that the remission of the diabetes is due to the direct effect of the operation more that the secondary effect of the weight loss. The reason for the major effect on the glucose metabolism after gastric bypass surgery is still unaccounted for.

This PhD. project will try to unveil some of the mechanisms that could explain the effect of gastric bypass surgery on the glucose metabolism seen in patients with type 2 diabetes.

The hypothesis of the study is that a factor "X" will course the remission of the diabetes. This factor "X" is related to the anatomic changes of the gastro intestinal tract, by eliminating the foods passage through the distal part of the ventricle and the duodenum, in combination with the Roux- en-Y sling.

The PhD. project will consist of clinical trails on patients that will undergo gastric bypass surgery. The studies will take place before and within the 1. week after surgery. The investigators will measure different hormones and adipokines in fast and the postprandial state. To discover possible new proteins the investigators will run proteomic on some samples. All the results will be compared to the same parameter on patients undergoing gastric banding, where the anatomy of the intestine hasn't been changed.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria in Denmark for undergoing gastric bypass and see the above study and cohort description.
* Well treated hypertension < 145/85. HbA1C <8,5 % and c-peptid> 700pmol/l

Exclusion Criteria:

* In treatment with antidepressive, DPP-4 inhibitors and intreatment for thyroid problems.
* Patients treated with insulin.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patiens undergoing gastric bypass surgery with or without type 2 diabetes and patients with diabetes undergoing gastric banding
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2009-01; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
What is the factor "X" that cause the remission of type 2 diabetes after gastric bypass | about 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Hvidovre Hospital, Hvidovre, Denmark

REFERENCES:
- [Derived] Palleja A, Kashani A, Allin KH, Nielsen T, Zhang C, Li Y, Brach T, Liang S, Feng Q, Jorgensen NB, Bojsen-Moller KN, Dirksen C, Burgdorf KS, Holst JJ, Madsbad S, Wang J, Pedersen O, Hansen T, Arumugam M. Roux-en-Y gastric bypass surgery of morbidly obese patients induces swift and persistent changes of the individual gut microbiota. Genome Med. 2016 Jun 15;8(1):67. doi: 10.1186/s13073-016-0312-1. PMID 27306058
- [Derived] Jorgensen NB, Dirksen C, Bojsen-Moller KN, Kristiansen VB, Wulff BS, Rainteau D, Humbert L, Rehfeld JF, Holst JJ, Madsbad S, Clausen TR. Improvements in glucose metabolism early after gastric bypass surgery are not explained by increases in total bile acids and fibroblast growth factor 19 concentrations. J Clin Endocrinol Metab. 2015 Mar;100(3):E396-406. doi: 10.1210/jc.2014-1658. Epub 2014 Dec 23. PMID 25536209
- [Derived] Jorgensen NB, Jacobsen SH, Dirksen C, Bojsen-Moller KN, Naver L, Hvolris L, Clausen TR, Wulff BS, Worm D, Lindqvist Hansen D, Madsbad S, Holst JJ. Acute and long-term effects of Roux-en-Y gastric bypass on glucose metabolism in subjects with Type 2 diabetes and normal glucose tolerance. Am J Physiol Endocrinol Metab. 2012 Jul 1;303(1):E122-31. doi: 10.1152/ajpendo.00073.2012. Epub 2012 Apr 24. PMID 22535748